CLINICAL TRIAL: NCT05884723
Title: Implementation of a Preoperative Ketogenic Diet for Reduction of Hepatic Steatosis Prior to Hepatectomy: a Randomized Control Trial
Brief Title: Preoperative Ketogenic Diet for Reduction of Hepatic Steatosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122435
Record Dates: First submitted 2023-05-15; First posted 2023-06-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Liver Steatoses; Liver Metastasis Colon Cancer; NAFLD
Keywords: ketogenic diet; NAFLD; colorectal liver metastases
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: preoperative ketogenic diet group vs control standard of care preoperative diet
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The surgeons, surgical team, and data abstractors will be blinded to participant randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet Arm (Experimental): Participants in this group will be counselled by a registered dietician and then undergo a 4-week preoperative well formulated ketogenic diet. They will record all nutritional uptake during the diet using an app called Cronometer and provide weekly summary reports to the study team.
  Interventions: Dietary Supplement: Ketogenic Diet
- Control Arm (No Intervention): Participants in this group will be counselled by a registered dietician and then undergo a 4-week standard of care diet, as recommended by Canada's Food Guide. They will record all nutritional uptake during the diet using an app called Cronometer and provide weekly summary reports to the study team.

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — 4-week preoperative well-formulated very low carbohydrate isocaloric diet consisting of 50g net daily carbohydrates and 1.5g/kg protein with the remaining energy needs consisting of primarily mono- and polyunsaturated fats
  Arms: Ketogenic Diet Arm

SUMMARY:
Non-alcoholic fatty liver disease is becoming increasingly common in Canada and throughout the world. Fatty liver can increase the risks of perioperative complications for those who need liver surgery. A ketogenic diet is low in carbohydrates and can be very effective in reducing liver fat content. The purpose of this randomized control trial is to compare the effect of a short duration (4 week) preoperative ketogenic diet on operative and disease outcomes in patients undergoing liver surgery. One arm will be randomized to the ketogenic diet and the other will receive standard of care pre-operative dietary consultation.

DETAILED DESCRIPTION:
The rise in obesity has contributed to increasing rates of non-alcoholic fatty liver disease (NAFLD) in Canada and globally. In the setting of liver surgery, fatty liver has been associated with higher rates of blood loss during surgery as well as higher rates of postoperative complications. A pre-operative ketogenic diet (KD) has been proposed as a strategy to decrease the risks of fatty liver in patients undergoing liver surgery and has shown promising results in reducing liver fat content, even with short-duration diets. The current literature contains a large variety of pre-operative diets aimed at reducing liver fat content and most studies are observational. Presently, there is no randomized control trial looking at the effects of a well-formulated and standardized KD prior to liver surgery and its effect on operative and disease outcomes. This study will randomize patients with NAFLD needing surgery to remove liver tumors to either the control group or intervention group. Patients in the control group will receive dietary consultation for a standard of care diet as recommended by Canada's Food Guide. Patients in the intervention group will consult with a dietician before starting a 4-week preoperative well-formulated very low carbohydrate KD. All participants will track daily nutritional intake and provide weekly summary reports via an app called Cronometer. The investigators will analyze differences in intraoperative blood loss and OR time, postoperative complications, disease recurrence and mortality rates between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older undergoing any type of liver resection (e.g. wedge, formal hepatectomy), either open or laparoscopic, for colorectal liver metastases (CRLM)
* Patients with evidence of hepatic steatosis on pre-operative imaging (CT or MR) or biopsy.
* Ability to use an app based nutritional program to track macronutrient uptake throughout the dietary intervention.

Exclusion Criteria:

* Patients undergoing liver resection for any other indication
* Patients on sodium glucose co-transporter 2 (SGLT-2) inhibitors (these are contraindicated with a ketogenic diet).
* Patients without evidence of hepatic steatosis.
* Patients with evidence of liver fibrosis or cirrhosis on preoperative bloodwork or imaging.
* Patients with alcohol-related hepatic steatosis.
* Patients with a known bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood transfusion | postoperative days 0-7
  receipt (binary) of packed red blood cell (pRBC) units intraoperatively and during the immediate postoperative time period (POD 0 - 7)

SECONDARY OUTCOMES:
Amount of perioperative blood transfusion | postoperative days 0-7
  Number of pRBC units transfused
Intraoperative blood loss | Operative period
  Intraoperative blood loss: measured by net sponge weight and fluid suctioned minus irrigation fluid
Steatosis | Time of primary surgery
  Level of steatosis in liver resection specimen
Change in steatosis | ~6 weeks
  Change in steatosis in liver pre-diet vs day of surgery
Operative time | During primary surgery
  time from surgery start to surgery stop
Postoperative complications | Postoperative days 0-30
  Postoperative complications (measured via the Clavien-Dindo Index) will be assessed within 30 days of the operation.
Postoperative length of hospital stay | Postoperative days 0-30
  Postoperative length of hospital stay will be assessed.
Postoperative hospital readmission | Postoperative days 0-30
  Hospital readmission will be assessed within 30 days of the operation
Postoperative rates of reoperation | Postoperative days 0-30
  Reoperation rates will be assessed within 30 days of the initial surgery.
Postoperative liver failure | Postoperative days 0-30
  Liver failure rates will be assessed within 30 days of the initial surgery.
Postoperative mortality | Postoperative days 0-30
  Mortality rates will be assessed within 30 days of the initial surgery.
Adherence to ketogenic diet | 4 weeks
  whether participants adhered to the diet assigned to them
Disease recurrence | 0 - 5 years postoperatively
  Time to disease recurrence will be assessed up to 5 years postoperatively.
Measurement of circulating cell-free tumor DNA | 0 - 5 years postoperatively
  Circulating cell-free tumour DNA levels will be measured up to 5 years postoperatively.
Cancer-related mortality | 0 - 5 years postoperatively
  Cancer-related mortality rates will be assessed up to 5 years postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Skaro, MD PhD, Principal Investigator — London Health Sciences Centre/Lawson Health Research Institute

IPD SHARING:
Plan to Share IPD: No